CLINICAL TRIAL: NCT06890455
Title: Fecal Calprotectin in Patients Infected with Intestinal Protozoan Infections
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Youstina Kamel Boles, Demonstrator of Medical parasitology, Sohag University
Other Study IDs: Soh-Med--25-3-07MS
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Fecal Calprotectin in Intestinal Protozoa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Case group: 40 patients complaining of gastrointestinal manifestations and infected with Blastocystis or Entamoeba histolytica
- Control group 1: 40 persons complaining of gastrointestinal manifestations without any protozoal infections
- Control group 2: - 40 healthy control cross-matched volunteers (without gastrointestinal manifestations, or intestinal parasites).

SUMMARY:
Calprotectin extracted from stool can be detected easily using ELISA. Numerous studies have shown that fecal calprotectin concentrations demonstrate a good correlation with intestinal inflammation This study aims to detect the relationship between fecal calprotectin and Blastocystis hominis and Entamoeba histolytica infections.

ELIGIBILITY:
Inclusion Criteria:

120 fecal samples will be collected as the following:

* 40 samples from patients complaining of gastrointestinal manifestations and only infected with B.hominis and E.histolytica.
* 40 samples from patients complaining of gastrointestinal manifestations without any protozoal infection.
* 40 healthy control cross-matched volunteers (without gastrointestinal manifestations, or intestinal parasites).

Exclusion Criteria:

* persons received antiparasitic drugs or antibiotic 2 weeks before sample collection Patients with mixed intestinal protozoa Patients with intestinal protozoa rather than Entamoeba histolytica and Blastocystis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 120 fecal samples will be collected as the following:
  * 40 samples from patients complaining of gastrointestinal manifestations and only infected with B.hominis and E.histolytica.
  * 40 samples from patients complaining of gastrointestinal manifestations without any protozoal infection.
  * 40 healthy control cross-matched volunteers (without gastrointestinal manifestations, or intestinal parasites).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Blastocystis and Entamoeba | 2 months

SECONDARY OUTCOMES:
Number of persons have high fecal calprotectin | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet